CLINICAL TRIAL: NCT04414462
Title: Comparison of Exergaming and Vestibular Training on Gaze Stability, Balance and Gait Performance of Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/00743 Amina bukhari
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Older Adults
Keywords: Exergaming; vestibular training; gaze stability; Balance; Gait; older adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Group I will receive following exergaming training: heading, tightrope tension,snowboard slalom and table tilt game
  Interventions: Other: exergaming training
- Group II (Active Comparator): Group II will receive Habituation,wobble board exercises,double leg,single leg and tandem stance training.
  Interventions: Other: training - Group II

INTERVENTIONS:
Other: exergaming training — * HEADING: For 5 mins a day,3 days a week in first 3 weeks (beginner level game) and for 10 mins a day, 3 days a week for 3 weeks. (advanced level game)
  * TIGHTROPE TENSION: For 5 mins a day,3 days a week in first 3 weeks (beginner level game) and for 10 mins a day, 3 days a week for 3 weeks. (advanced level game)
  * SNOWBOARD SLALOM: For 5 mins a day,3 days a week in first 3 weeks (beginner level game) and for 10 mins a day, 3 days a week for 3 weeks. (advanced level game)
  * TABLE TILT: For 5 mins a day,3 days a week in first 3 weeks (beginner level game) and for 10 mins a day, 3 days a week for 3 weeks. (advanced level game)
  Arms: Group I
Other: training - Group II — * Wobble board for 4 mins a day,3 days a week for first 3 weeks and for 8 mins a day,3 days a week for 3 weeks.
  * Habituation exercises for 4 mins a day,3 days a week for first 3 weeks and for 8 mins a day,3 days a week for 3 weeks.
  * Double leg stance with eyes open and eyes closed on firm surface and on foam for 4 mins a day,3 days a week for first 3 weeks and for 8 mins a day,3 days a week for 3 weeks.
  * Single leg stance with eyes open and eyes open on firm surface and on foam for 4 mins a day,3 days a week for first 3 weeks and for 8 mins a day,3 days a week for 3 weeks.
  * Tandem walk stance with eyes open and eyes closed on firm surface and on foam for 4 mins a day,3 days a week for first 3 weeks and for 8 mins a day,3 days a week for 3 weeks.
  Arms: Group II

SUMMARY:
Exergames showed beneficial effects than conventional exercises for gaze stability, balance and gait improvements in older individuals. Further studies should be conducted to explore the benefits of exergames on older adults. This study aims to explore that exergaming has more effects on gaze stability, balance and gait performance of older individuals.

DETAILED DESCRIPTION:
According to a recent report by 2050, the global adult population between the age 65 and above is expected to increase to 28%. A total of 12.13 million people in Pakistan are above age of 60, which is expected to raise to 17.53 million by 2025. A high quality of life as well as longevity is considered important in older adults.However, characteristics of aging include a decrease in muscle strength, balance and decreased vestibular functions can lead to falls and compromise good health in older adults.

Vestibular rehabilitation is an exercised based program intended to alleviate both primary and secondary problems caused by vestibular disorders.The main focus of vestibular rehabilitation is to use the existing vestibular system for gaze, postural stability and gait by use of somatosensory and visual cues. Depending on the vestibular disorders three main types of exercises are used. Habituation Gaze stability exercises ,Balance training. Habituation exercises are indicated for patients who complain of dizziness during quick head movements and when they change position like when they bend over or look up to reach above their head. The goal of habituation exercise is to reduce the dizziness through repeated exposure to specific movements or visual stimuli that provoke patient's dizziness.

Gaze stability exercises include eyeball movement, saccadic eye movement, pursuit eye movement, vergence eye movement, vestibular-ocular reflex exercise. These exercises improve the static balance control thus improves postural control required for vestibular function and can be mediated by VSR improvements. These exercises are useful in bilateral vestibular hypofunction. Balance training are used to improve standing, bending, reaching and performance of dual tasks on even and uneven surfaces. These exercises proved to be effective in making individuals do activities of daily livings and prevents the risks of falls.

Computer based technology is becoming popular in rehabilitation. It stimulates learning in real-life environment and provides a 3-dimensional sensory feedback. A computer-generated technology allows the user to interact with a virtual world and to make correction during performing an exercise task. In particular, previous studies have suggested that new technology, such as the Wii Fit Board (WFB) can be used for balance training using virtual reality These games have showed repeated good results in vestibular rehabilitation of elderly.Virtual reality enables the individual to be physically active and provides a pleasant and motivating way of training in these individuals.

There are literature for the safe and effective use of exergaming in improving gaze stability, balance and postural control in older individuals Jaap Swanenburg et al concluded that exergaming is effective in improving gaze stability, balance and postural control in older adults .Lynne M Taylor showed that active video games proved to be effective in improving balance and gait in older individuals .J Hashim concluded that Exergames improved dynamic balance in older adults when compared with conventional exercises.

ELIGIBILITY:
Inclusion Criteria:

* A score of 21 and above on berg balance scale.
* A minimum head velocity of 150◦/s on dynamic visual acuity test.

Exclusion Criteria:

* Acute Musculoskeletal pain
* Uncontrollable cardiovascular disease (e.g. High blood pressure, Uncontrolled sugar)
* Weakness from known neurological problems (Parkinson's, stroke, multiple sclerosis)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test (TUG) | Change from Baseline balance to 6th Weeks
  TUG is a test used to assess a person's mobility. TUG measured the time required for an individual to stand up from a chair with armrests, walk 3 m, turn, walk back to the chair, and sit down. Normal healthy elderly usually completes the task in ten seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more.
Dynamic Visual Acuity | Change from Baseline vestibular ocular reflex to 6th Week
  It provides an objective and instrumented way of assessing Vestibulo-ocular reflex (VOR)function in response to rotational and functional head movement stimuli. The DVA testing system consisted of a personal computer with a monitor and a velocity sensor which is fixed on a headset to the participant's head. Minimum acceptable head testing velocity was 150◦/s.
Dynamic Gait Index | Change from Baseline gait to 6th Week
  Dynamic gait index is used to assess gait, balance and fall risk. It is a valuable clinical tool for evaluating dynamic balance in community dwelling older adults. Total score is 24, a score < 19/24 is predictive of falls risk in community dwelling elderly

SECONDARY OUTCOMES:
Force Platform | Change from Baseline postural variation to 6th Week
  It provides a quantitative way to measure postural control and analysis of various aspects of balance.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Pakistan General Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomita Y, Arima K, Tsujimoto R, Kawashiri SY, Nishimura T, Mizukami S, Okabe T, Tanaka N, Honda Y, Izutsu K, Yamamoto N, Ohmachi I, Kanagae M, Abe Y, Aoyagi K. Prevalence of fear of falling and associated factors among Japanese community-dwelling older adults. Medicine (Baltimore). 2018 Jan;97(4):e9721. doi: 10.1097/MD.0000000000009721. PMID 29369207
- [Background] Siddiqi FA, Masood T, Osama M, Azim ME, Babur MN. Common balance measures and fall risk scores among older adults in Pakistan: Normative values and correlation. J Pak Med Assoc. 2019 Feb;69(2):246-249. PMID 30804593
- [Background] Lee Y, Choi W, Lee K, Song C, Lee S. Virtual Reality Training With Three-Dimensional Video Games Improves Postural Balance and Lower Extremity Strength in Community-Dwelling Older Adults. J Aging Phys Act. 2017 Oct 1;25(4):621-627. doi: 10.1123/japa.2015-0271. Epub 2017 Sep 19. PMID 28290746
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Treatment for Vestibular Disorders: How Does Your Physical Therapist Treat Dizziness Related to Vestibular Problems? J Neurol Phys Ther. 2016 Apr;40(2):156. doi: 10.1097/01.NPT.0000481898.55592.6e. No abstract available. PMID 26934418
- [Background] Swanenburg J, Babler E, Adelsberger R, Straumann D, de Bruin ED. Patients with chronic peripheral vestibular hypofunction compared to healthy subjects exhibit differences in gaze and gait behaviour when walking on stairs and ramps. PLoS One. 2017 Dec 18;12(12):e0189037. doi: 10.1371/journal.pone.0189037. eCollection 2017. PMID 29253883
- [Derived] Bukhari SA, Ghous M, Butt P, Kiyani SK, Tariq A. Comparison of exergaming and vestibular training on gaze stability, balance, and gait performance of older adults: A single blind randomized control trial. J Pak Med Assoc. 2022 Oct;72(10):1909-1912. doi: 10.47391/JPMA.3566. PMID 36660969